CLINICAL TRIAL: NCT00353275
Title: Studies on Hyperglycemia in Surgical Infections
Brief Title: Hyperglycemia in Surgical Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling eligible patients
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Lillian Kao, Professor - Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-04-209; 1K23RR020020-01A1 (NIH)
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Necrotizing Fasciitis
Keywords: Strict glycemic control
MeSH Terms: conditions — Fasciitis, Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Strict glycemic control with a blood glucose target range of 80-110 mg/dL
  Interventions: Drug: Strict Glycemic control
- 2 (Other): Conventional glycemic control with blood glucose target range of 110-140 mg/dL
  Interventions: Drug: Conventional Glycemic Control

INTERVENTIONS:
Drug: Strict Glycemic control — Blood glucose target range is 80-110 mg/dL.
  Arms: 1
Drug: Conventional Glycemic Control — Blood glucose target range is 110-140 mg/dL.
  Arms: 2

SUMMARY:
The primary purpose of this study is to evaluate two glycemic control regimens on clinical outcome in patients with necrotizing soft tissue infections. Secondary aim is to evaluate the inflammatory and immune responses to the glycemic control regimens.

DETAILED DESCRIPTION:
This is a multi-center explanatory trial of strict glycemic control for surgical patients with necrotizing soft tissue infection (NSTI). The primary objective of this study is to verify feasibility of the intervention, provide unbiased and evidence-based estimates of treatment effects, and obtain data needed to design and direct a larger multi-center trial if necessary. The multi-center trial (n >100) will have adequate power to identify a 30% difference in favorable outcome defined as discharge alive from the hospital without an amputation in less than the median number of hospital days. Secondary objectives include evaluation of specific hypotheses relating the intervention to cytokine and neutrophil responses. These preliminary data will provide the basis for future research and grant applications, lend insight into the mechanisms by which hyperglycemia results in adverse effects, and improve outcome through the development of evidence-based therapeutic strategies for patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be enrolled at one of the following centers: the LBJ General Hospital (UT-Houston), the Ben Taub General Hospital (Baylor Houston), The Methodist Hospital (Texas Medical Center), or the University of Texas Health Science Center at San Antonio and the Brooke Army Medical Center.
* We will attempt to enroll all eligible patients with a diagnosis of a necrotizing soft tissue infection (NSTI), including Fournier's gangrene, confirmed in the operating room regardless of age, ethnicity or gender.

Exclusion Criteria:

* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian S Kao, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - LBJ General Hospital/ UT health Science Center-Houston, Houston, Texas
  - Brooke Army Medical Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11) | 59 (5) | 59 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
Weight [Mean (Full Range); unit: pounds] | 169 [158 to 180] | 240 [215 to 272] | 212 [158 to 272]
Height [Mean (Full Range); unit: inches] | 66 [65 to 67] | 65 [63 to 68] | 66 [63 to 68]

OUTCOME MEASURES:

1. Primary Outcome: Infectious Morbidity
Time Frame: Duration of hospital stay, an average of 2 weeks
Population: The study was stopped because it appeared we would not be able to enroll enough patients into the study by the time funding would conclude. Because only a total of 5 patients were enrolled and underwent study procedures, there was not enough data to be analyzed.
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Composite Outcome (Favorable Outcome Defined as Discharge Home, Without an Amputation, in Less Than the Median Hospital Stay for Survivors)
Time Frame: Duration of hospital stay
Population: as for outcome 1
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Organ Failure
Time Frame: Duration of hospital stay
Population: as for outcome 1
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hypoglycemia
Time Frame: Duration of hospital stay
Population: as for outcome 1
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Strict Glycemic Control | Conventional Glycemic Control
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No